CLINICAL TRIAL: NCT05546580
Title: An Escalation/Expansion, Open Label, Multicenter Study of Iadademstat and Gilteritinib in Patients With Relapsed or Refractory Acute Myeloid Leukemia (R/R AML) With FMS-like Tyrosine Kinase Mutation (FLT3 Mut+): The FRIDA Study
Brief Title: Study of Iadademstat and Gilteritinib in Patients With R/R AML With FMS-like Tyrosine Kinase Mutation (FLT3 Mut+)
Acronym: FRIDA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oryzon Genomics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL04-ORY-1001
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
Keywords: Acute Myeloid Leukemia, FLT3 mut
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — iadademstat; gilteritinib

STUDY DESIGN:
Intervention Model Description: Escalation/extension open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active arm (Experimental): iadademstat and gilteritinib
  Interventions: Drug: Iadademstat; Drug: Gilteritinib Oral Tablet

INTERVENTIONS:
Drug: Iadademstat — iadademstat oral solution
  Other Names: ORY-1001, RO7051790
Drug: Gilteritinib Oral Tablet — 120 mg Gilteritinib
  Other Names: XOSPATA®

SUMMARY:
Iadademstat is being studied as a treatment for subjects with Relapsed or Refractory Acute Myeloid Leukemia (R/R AML) with FMS-like tyrosine kinase mutation (FLT3 mut+). During the trial, iadademstat will be given in combination with gilteritinib, a drug that is already approved to treat patients with FLT3-mutated R/R AML.

DETAILED DESCRIPTION:
This is an escalation/expansion, open label, single arm, study to investigate the safety and the RP2D of the combination of iadademstat with gilteritinib in FLT3-mutated R/R AML.

This study consists of 2 parts. A dose finding part to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) and emerging activity of iadademstat and gilteritinib combination, and to determine the pharmacologically-active dose (i.e., the minimum safe and biologically active dose) of iadademstat in combination with gilteritinib, and an expansion part at the specific dose/s selected to evaluate the activity of iadademstat in combination with gilteritinib in patients with FLT3-mutated R/R AML.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of primary AML or AML with myelodysplasia-related changes (AML-MRC)
* Patient is in first or second relapse or has refractory disease. Patients must have had histologic verification of AML at the original diagnosis.
* Patient must be positive for the following FLT3 mutations in bone marrow or PB: FLT3 internal tandem duplication (ITD), FLT3 tyrosine kinase domain (TKD) D835 or I836 or FLT3-ITD and specified FLT3-TKD.
* ECOG performance status 0-2
* Life expectancy of at least 3 months in the opinion of the investigator.
* Normal hepatic and renal function.
* Patient is able to swallow oral medications.
* Female patients are postmenopausal, documented as surgically sterile, use two methods of contraception or practice true abstinence and have a negative urine pregnancy test at screening.
* Male patients even if surgically sterilized agree to practice true abstinence or use highly effective barrier contraception.

Main Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia.
* Known BCR-ABL-positive leukemia.
* AML secondary to prior chemotherapy for other neoplasms (except for MDS).
* AML that has relapsed after or is refractory to more than 2 lines of therapy.
* Clinically active central nervous system leukemia or prior history of NCI CTCAE Grade ≥ 3 drug-related CNS toxicity.
* Major surgery or radiation therapy within 4 weeks prior to the first study dose.
* Prior treatment with iadademstat is not allowed. Treatment with any other agents with KDM1A/LSD1 inhibitory activity is only allowed if treatment finalized at least 3 weeks prior to first dose on study. Previous treatment with FLT3 inhibitors is allowed in the following cases: midostaurin and sorafenib are allowed when used in first-line therapy regimen as part of induction, consolidation and/or maintenance: quizartinib and gilteritinib are allowed when used in first-line therapy regimen, as part of induction, consolidation and/or maintenance, ONLY if patients were not refractory to the drugs or if responding, relapse did not occur while on these drugs.
* Patients not eligible to receive gilteritinib per label.
* Prior treatment with 3 or more lines of AML therapy.
* Treatment with any investigational products within 3 weeks prior to first dose of study treatment.
* Uncontrolled hypertension or poorly controlled diabetes.
* Evidence of active uncontrolled viral, bacterial, or systemic fungal infection.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | Up to 18 months
  Number of participants with Adverse Events (AE) after treatment with iadademstat in combination with gilteritinib in patients with FLT3-mutated R/R AML.
Laboratory value abnormalities and/or adverse events (AE) | Up to 18 months
  Number of participants with laboratory value abnormalities and/or Adverse Events (AE) after treatment with iadademstat in combination with gilteritinib in patients with FLT3-mutated R/R AML.
Vital sign abnormalities and/or adverse events (AEs) | Up to 18 months
  Number of participants with vital signs abnormalities and/or Adverse Events (AE) after treatment with iadademstat in combination with gilteritinib in patients with FLT3-mutated R/R AML.
Routine 12-lead electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to 18 months
  Number of participants with Routine 12-lead electrocardiogram (ECG )abnormalities and/or Adverse Events (AE) after treatment with iadademstat in combination with gilteritinib in patients with FLT3-mutated R/R AML.
Recommend Phase 2 dose (RP2D) | Up to 18 months
  Determine the recommended Phase 2 dose (RP2D) of iadademstat in combination with gilteritinib in patients with FLT3-mutated R/R
iadademstat tmax | Up to 26 days
  Measurement of the time it takes for iadademstat to reach the maximum concentration (Cmax) in blood.
Iadademstat Cmax | Up to 26 days
  Measurement of the highest concentration of iadademstat in the blood after a dose is given.
iadademstat Cmin | Up to 26 days
  Measurement of the lowest concentration of iadademstat in the blood, after a dose is given.
iadademstat AUC | Up to 26 days
  Measurement of how much iadadmestat reaches a person's bloodstream in a given period of time after a dose is given.
iadademstat Target Engagement (TE) | Up to 26 days
  Percent of drug covalently bound to LSD1 molecule
OR rate | Up to 18 months
  Proportion of patients achieving complete remission (CR), CR with incomplete hematologic recovery (CRi), and partial remission (PR).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 24 months
  Time from start of treatment to the time of death from any cause.
Event-Free-Survival (EFS) | Up to 18 months
  Time from start of treatment to the date of failure to achieve CR or CRi, relapse from CR/CRi, or death from any cause, whichever occurs first.
Overall response rate | Up to 6 months
  Percentage of patients with complete remission (CR), CR with incomplete blood count recovery (CRi), or PR.
Time to Response (TTR) | Up to 6 months
  Time from the date of initial dosing at RP2D/expansion dose to first documentation of either a type of CR or Partial Response (PR).
Duration of Remission (DoR) | Up to 18 months
  Time from the date of first documentation of any type of remission to the date of first documentation of progression of remission for remitters
Transfusion independence rate | Up to 18 months
  A patient is defined as red blood cell (RBC) and/or platelet-transfusion independent if he/she receives no RBC and/or platelet transfusions for a period of at least 8 weeks. Rate of transfusion independence is the percentage of patients who become RBC and/or platelet transfusion independent (from the number of patients transfusion dependent at baseline).
Transplantation Rate Time Frame | Up to 18 months
  Percentage of patients undergoing Hematopoietic Stem Cell Transplantation (HSCT) during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Reale-Vidal, MD, Study Chair — Oryzon Genomics
Locations (13):
- United States (13):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - The John Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Rutgers, The State University, Piscataway, New Jersey
  - Icahn School of Medicine at Mount Sinai and Mount Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee
  - West Virginia University, Morgantown, West Virginia
  - Froedtert Hospital & The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No